CLINICAL TRIAL: NCT05404399
Title: A Randomised Control Trial Evaluating the Use of a Combined Preformulated Exercise Plan in the Improvement of Musculoskeletal Health in Patients With Generalised Neck and Low Back Pain.
Brief Title: Free From Pain Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP0629
Record Dates: First submitted 2022-05-27; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-02

CONDITIONS: Musculoskeletal Pain; Quality of Life; Fear of Falling
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free From Pain Exercise Book (Experimental): Participants in Group 1 will be asked to engage in the 3 sets of exercises within the exercise book for the following 12 weeks. They will be advised to engage in the exercises at least five times a week. The ideal plan would be as follows:
  Monday - Otago exercises. Tuesday - Neck and Back exercises. Wednesday - Otago exercises. Thursday - Reading the weekly reading material. Friday - Neck and Back exercises. Saturday - Otago exercises. Sunday - Rest day.
  Furthermore, it will be recommended that participants in Group 1 read one motivation/reason chapter and one metaphor each week for 12 weeks, to ensure that they absorb the information fully and do not overbear themselves with information.
  Participants in Group 1 will also be asked to fill in the exercise diary, found at the back of the exercise book, each time they exercise as part of the "Free From Pain" programme.
  Interventions: Behavioral: "Free From Pain Exercise Book"
- Usual Care (physiotherapy) (Active Comparator): Those in Group 2 (control group) will not be provided with the "Free From Pain Exercise Book", and will instead be referred to physiotherapy as part of standard / usual care. They will be asked to report when their physiotherapy commenced.
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: "Free From Pain Exercise Book" — Participants in Group 1 will be provided with the "Free From Pain Exercise Book".
  Arms: Free From Pain Exercise Book
Behavioral: Physiotherapy — Participants in Group 2 would be referred to Physiotherapy (usual care)
  Arms: Usual Care (physiotherapy)

SUMMARY:
To determine the effectiveness of the "Free From Pain" Exercise Book containing the preformulated 12-week "Free From Pain" exercise programme in reducing pain, improving quality of life and decreasing fear of falling in people over 60 years of age when compared to usual care (referral to physiotherapy).

DETAILED DESCRIPTION:
According to the World Health Organisation, over 1.5 billion people have musculoskeletal conditions worldwide. Musculoskeletal conditions can cause significant pain, leading to extended periods of immobility and subsequent disability. This causes a loss of fitness, increasing the threat of conditions associated with inactivity, such as cancer and cardiovascular disease. Inactivity will also reduce muscle mass, bringing an increased risk of falls and fall-related injuries. Fortunately, exercise can bring about many health benefits in older age, by improving functional ability and well-being. Additionally, specific programmes which focus on balance and strength reduce the risk and rate of falls. Currently, the most popular rehabilitation modality for seniors is physiotherapy. Unfortunately, there is a huge demand for physiotherapy and there is a waiting period. Waiting for physiotherapy services may have detrimental effects on pain, disability, quality of life, and psychological symptoms in persons with musculoskeletal disorders. A more inexpensive and readily available intervention could therefore be desirable to manage musculoskeletal pain in seniors.

The "Free from Pain" exercise programme, found within the "Free From Pain" exercise book, is a fusion of three different generally accepted exercise programmes. The three programmes are the Otago exercises for lower body strength and balance, the motor control exercises for the lower back and the isometric exercises for the neck and shoulder. Developed by Robertson and Campbell for the New Zealand Accident Compensation Corporation (ACC), the Otago exercise programme aimed to improve balance and strength in patients in order to prevent falls. As a secondary effect, the Otago exercise programme also reduces musculoskeletal pain in community-dwelling older adults. Along with the exercises, the "Free From Pain Exercise Book" also contains 13 chapters. These comprise an introductory chapter, 12 motivation/reason to exercise chapters and 12 exercise-related metaphors.

This is a randomised control trial that will be conducted over a 12-week period. The study population will include 60 participants who will be randomised into a test group and a control group. Participants in the test group (Group 1) will be provided with the "Free From Pain Exercise Book" and participants in the control group (Group 2) would be referred to Physiotherapy (usual care). Participants in the test group (Group 1) will be asked to engage in the 3 sets of exercises within the exercise book for the following 12 weeks. They will be advised to engage in the exercises at least five times a week, whilst reading the informative material once a week. Participants will be asked to provide data in the form of completed surveys at the beginning and the end of the study period.

The aim of the study is to investigate whether the "Free From Pain" exercise Book, containing the preformulated 12-week exercise programme, reduces pain, improves quality of life and decreases fear of falling in people over 60 years of age more than usual care (referral to physiotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 60 years of age.
* Have generalised neck, low back and/or musculoskeletal pain.
* Clinical patient not requiring surgical intervention or patient not keen on surgical intervention

Exclusion Criteria:

* Lacking the physical ability or cardiovascular fitness required to participate in an exercise programme. This criterion will be explained on the participant information sheet by stating: "If you are unable to walk up a flight of stairs without getting breathless, please do not apply for participation in this study".
* Self-identified lack of mental ability to participate in the exercise programme.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in musculoskeletal health as assessed by the Musculoskeletal Health Questionnaire (MSK-HQ) | Baseline and 12 weeks
  The Musculoskeletal Health Questionnaire (MSKHQ), developed by Arthritis Research UK, has been shown to be an easy to understand and relevant survey that is widely used in musculoskeletal health research. For this outcome measure, the minimal clinical difference is a change of 6 points or more in the participant's score.

SECONDARY OUTCOMES:
Changes in musculoskeletal health as assessed by a Visual Anlogue Scale (VAS) | Baseline and 12 weeks
  Improvements in 10-point VAS scale for perceived musculoskeletal pain in the lower back, hips, knees, ankles, and feet, where 0 denotes no pain and 10 denotes extremely severe pain. The Visual Analogue Scale (VAS) is a validated, subjective measure of acute and chronic pain.
Changes in health-related quality of life as assessed by the EuroQol- 5 Dimension (EQ-5D) | Baseline and 12 weeks
  Improvement in EQ-5D. The EuroQol- 5 Dimension (EQ-5D) questionnaire, first developed by the EuroQol Group, evaluates health-related quality of life in a simple survey.
Chanes in a fear of falling as assessed by the short Falls Efficacy Scale-International (short FES-I) | Baseline and 12 weeks
  Improvement in short FES-I. The short Falls Efficacy Scale-International (short FES-I) is a 7-item version of the FES-I. This version has been validated for community-dwelling older population. Furthermore, the short FES-I can predict future falls, muscle weakness, frailty, and overall disability.
Participant opinion on the reading mateiral provided as assessed by the Usefulness scale for patient educational material (USE) | 12 weeks
  Usefulness scale for patient educational material (USE) will be used to assess the usefulness of the information provided.
Participant compliance to the exercise programme as assessed by an exercise diary | 12 weeks
  Participant compliance to the exercise programme as assessed using the "Free From Pain" exercise diary for Group 1 participants in order to determine the effects of the programme with relation to intervention acceptance.
Length of physiotherapy treatment | 12 weeks
  Participants in Group 2 will be asked to provide the date when physiotherapy commenced.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool University Hospitals Nhs Foundation Trust, Liverpool, Merseyside, United Kingdom